CLINICAL TRIAL: NCT03936803
Title: Interval Training Versus Electro Acupuncture on Liver Functions in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ramy Salama Atia Draz, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001579
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Active Comparator): Twenty-five patients suffering from Nonalcoholic fatty liver disease (NAFLD) and taking their standard medications in addition to aerobic interval training exercise .Its consisted of cycle ergometer training, 3 days a week for 6 weeks. Aerobic interval training consisted of ( 8 )minutes warm-up, followed by 4 times of 4-minute intervals with heart rate (HR) at 85% of sub maximum HR, with active pauses of 3 minutes of walking at 60% of sub maximum heart rate HR. The exercise session was terminated by 5 minutes cool-down
  Interventions: Behavioral: aerobic interval training exercise .
- electro-acupuncture group (Active Comparator): Twenty-five patients suffering from Nonalcoholic fatty liver disease (NAFLD), and taking their standard medications In addition to electro acupuncture (EA) of (2 Hz, 4 mA) was applied at points of: liver 3 (LR3) ,liver 14 (LR14), gall bladder 34 (GB 34) and stomach 36 (ST36) .
  Duration of the session was 15 min / each, three sessions per week for six weeks
  Interventions: Device: electro acupuncture

INTERVENTIONS:
Behavioral: aerobic interval training exercise . — Its consisted of cycle ergometer training, 3 days a week for 6 weeks. Aerobic interval training consisted of ( 8 )minutes warm-up, followed by 4 times of 4-minute intervals with HR at 85% of sub maximum HR, with active pauses of 3 minutes of walking at 60% of sub maximum HR. The exercise session was terminated by 5 minutes cool-down
  Arms: exercise group
Device: electro acupuncture — electroacupuncture (EA) of (2 Hz, 4 mA) was applied at points of:liver 3 LR3,liver 14 LR 14, gall bladder 34 (GB 34) and stomach 36 (ST36) .
  Duration of the session was 15 min / each, three sessions per week for six weeks
  Arms: electro-acupuncture group

SUMMARY:
in this study, the investigators compare the effect of interval training exercise and electroacupuncture on liver functions in non-alcoholic fatty liver disease patients

DETAILED DESCRIPTION:
fifty patients suffering from Nonalcoholic fatty liver disease (NAFLD) will be recruited in this study with age ranged from 30-55 years old from both sexes, chosen from internal medicine department at Kasr El Aini hospital and from the outpatient clinic of nutrition and cardiovascular disorders at the faculty of Physical Therapy Cairo University, they were divided in to two groups:Group (1):

Twenty-five patients suffering from Nonalcoholic fatty liver disease (NAFLD), and taking their standard medications In addition to electroacupuncture at points of LR3 (Taichong), LR14 (Qimen), GB 34(Yanglingquan) and ST36 (Zu San Li). Group (2):

Twenty-five patients suffering from Nonalcoholic fatty liver disease(NAFLD) and taking their standard medications in addition to aerobic interval training exercise.Lab investigations of:

Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Triglycerides (TG) and C-reactive protein (CRP).to judge liver functions

ELIGIBILITY:
Inclusion Criteria:

1. Sixty patients suffering from Nonalcoholic fatty liver disease (NAFLD).
2. Their age will be ranged from 30-55 years old.
3. Body mass index (30 - 40)
4. All patients are medically stable.

Exclusion Criteria:

* Patients with Hepatitis C & b
* Acute and chronic significant illnesses that may interfere with actual training, severe ventricular arrhythmia, hemodynamic deterioration or exercise-induced arrhythmia at baseline testing.
* Co-morbidities that limit exercise tolerance (hemoglobin 10 g/dl, a chronic obstructive pulmonary disease with FEV1 50%).
* Hypertension (resting blood pressure >140/90 mmHg).
* Heart failure, inability to exercise, or drug abuse.
* Pacemakers
* Pregnancy
* Epileptic Seizures
* Cancer

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
body mass index | about 4 weeks
  was used for measuring the weight and height of each patient to calculate the body mass index (BMI) (figure). BMI = weight kg / (height m)2
lab investigations | about 12 weeks
  lab investigation of aminotransferase (ALT) iu/l and Aspartate aminotransferase (AST) iu/l There was a subjective evaluation of the level of exhaustion throw observation of ventilation, walking action and fascial expression in patients at the end stage of test.
  * Subjects initially performed submaximal exercise stress test (increasing 1 W every 2 s) on an electronically braked cycle ergometer to determine sub maximum heart rate.
lab investigations | about 14weeks
  lab investigation of Triglycerides (TG) mg/dl and c-reactive protein mg/l

CONTACTS AND LOCATIONS:
Overall Officials: zahra 63 serry, prof, Study Director — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt